## Informed consent for participation in a medical research project

Titel of the research project: A new intelligent stocking for quantification of edema in the lower limbs

## **Declaration from the participant:**

I have received both written and oral information and I know enough about the purpose, methods and pros and cons to accept participation.

I know <u>participation is volunteer</u> and I am always able to withdraw my consent without losing current or future rights for receiving treatment.

I hereby gives my consent to participate in the research project, and I confirm, that I received a copy of this document as well as copies of the written information of the project.

| Name of study participant: | |
|---|---|
| Date: | Signature: |
| | ng your health is discovered, you will be informed. If you <b>do not</b> want to your health discovered during this study, please mark it here: |
| Do you want to receive res | ults of the research project and possible consequences for you?: |
| Yes (write x) | No (write x) |
| Declaration from the inf | ormant: |
| I declare, that the participa | ant has received both oral and written information about the project. |
| From my perspective, I have whether you want to partic | ve been given enough information about the project, and you are able to judge ipate or not. |
| Name of the informant: | |
| Date: | Signature: |

Project identification: Version 1, marts 14, 2018.